CLINICAL TRIAL: NCT06426862
Title: To Determine the Effects of the Otago Exercise Program on the Frequency of Falls, Balance Capabilities, and Overall Physical Performance in Stroke Patients.
Brief Title: Effects of Otago Exercise Program in Falls, Balance and Physical Performance in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC 01741 Muhammad Baqir
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Stroke; Cardiovascular Attack; Otago Exercise Program; Berg Balance Scale; Time Up & Go Test; Fugl-Meyer Assessment
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): The interventional group will receive both treatment routine physiotherapy and the Otago exercise program (OEP). The OEP is the exercise designed for strength and balance to improve mobility, functional balance and walking. The exercises included in this protocol are 17: strength, balance and walking. The participants will receive this protocol with 10 repetitions while the interval between exercises will not be fixed; patients will be given ample time to relax and recuperate before beginning another exercise, 3 times a week for six weeks and the time duration will be 30 to 45 minutes. The exercises will be progressively administered weekly.
  Interventions: Other: Otago Exercise Program; Other: Control Group
- Control group (Active Comparator): The control group will receive routine treatment of physiotherapy for strokes like strengthening of upper and lower limb muscles (knee flexor, hip adductor and ankle dorsiflexor), stretching (hip abductors and ankle plantar flexor), postural awareness, gait and balance training like static and dynamic. The participants will be assessed through baseline assessment.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Otago Exercise Program — Otago exercise program
  Strengthening Exercise Knee extensor, Hip adductors, heel and toe raising
  Balance exercise Sit to stand, Knee bending, one leg standing, tandem stance, side walk, walk and turn around, tandem walk, backward walk, heel and toe walk, stair climbing
  Arms: Interventional Group
Other: Control Group — Routine physiotherapy like strengthening, stretching, postural awareness, gait and balance training.

SUMMARY:
This study aims to determine the effects of the Otago Exercise Program (OEP) on falls and balance as well as overall physical performance. Participants will be divided into two groups; control and intervention group. It is a week-long study, the participants will be assessed through the Berg Balance Scale (BBS), Time Up and Go (TUG) and Fugl-Meyer Assessment (FMA).

DETAILED DESCRIPTION:
The previous literature suggested that the Otago exercise showed significant improvement in terms of fall and balance. Most of the Studies were conducted on the elderly population but limited studies are available regarding stroke. This study will look at the effect of Otago exercise on stroke patients. The Otago exercise consists of 17 exercises; strengthening and balancing exercises. The participants will receive Otago exercise and routine physiotherapy treatment for six weeks. The participants will go through three assessments; Baseline Assessment, After 3 weeks assessment and final assessment. For association, a mixed method ANOVA test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke
* Medically stable patients with acute to subacute level of stroke recovery (< 6 month).
* Patients 40 plus age
* Berg balance scale <45 and >20 score
* TUG test scoring >20 sec

Exclusion Criteria:

* Participants having cognition problem or language barrier
* Physical disability (fracture or amputation) other than stroke
* Previous surgery 6 weeks
* Cardiovascular and pulmonary disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline
  The BBS was used to assess the quantitative measure of balance and fall risk among the older population through direct observation of their performance. The 14 items scale of total scoring 56 and each item has a scaling of 0 to 4. The scoring up to 0 to 20 represents impaired balance, 21 to 40 indicate acceptable while >40 represent good balance.
Berg Balance Scale | After 3 weeks
  The BBS was used to assess the quantitative measure of balance and fall risk among the older population through direct observation of their performance. The 14 items scale of total scoring 56 and each item has a scaling of 0 to 4. The scoring up to 0 to 20 represents impaired balance, 21 to 40 indicate acceptable while >40 represent good balance.
Berg Balance Scale | After 6 weeks
  The BBS was used to assess the quantitative measure of balance and fall risk among the older population through direct observation of their performance. The 14 items scale of total scoring 56 and each item has a scaling of 0 to 4. The scoring up to 0 to 20 represents impaired balance, 21 to 40 indicate acceptable while >40 represent good balance.
Time Up & Go Test | Baseline
  The TUG test was used to assess the functional mobility of the participants. The gait and balance maneuvers used in daily life are attributed to functional mobility. The participants were required to stand up, walk away through 3 meters or 10 feet and turn back to sit in the chair at starting. The individuals who cover the distance in >20 seconds are considered as dependent in their activities while those who complete the task in <20 sec indicate independence in ADLs.
Time Up & Go Test | After 3 weeks
  The TUG test was used to assess the functional mobility of the participants. The gait and balance maneuvers used in daily life are attributed to functional mobility. The participants were required to stand up, walk away through 3 meters or 10 feet and turn back to sit in the chair at starting. The individuals who cover the distance in >20 seconds are considered as dependent in their activities while those who complete the task in <20 sec indicate independence in ADLs.
Time Up & Go Test | After 6 weeks
  The TUG test was used to assess the functional mobility of the participants. The gait and balance maneuvers used in daily life are attributed to functional mobility. The participants were required to stand up, walk away through 3 meters or 10 feet and turn back to sit in the chair at starting. The individuals who cover the distance in >20 seconds are considered as dependent in their activities while those who complete the task in <20 sec indicate independence in ADLs.
Fugl-Meyer Assessment | Baseline
  Motor impairment is the most common complication of stroke; it was measured by FMA quantitatively. The scale is divided into 5 domains; sensory & motor function, balance, joint range of motion and joint pain. Each domain has a scale of 0 to 2 score while the total scoring of the scale is 226 score.
Fugl-Meyer Assessment | After 3 weeks
  Motor impairment is the most common complication of stroke; it was measured by FMA quantitatively. The scale is divided into 5 domains; sensory & motor function, balance, joint range of motion and joint pain. Each domain has a scale of 0 to 2 score while the total scoring of the scale is 226 score.
Fugl-Meyer Assessment | After 6 weeks
  Motor impairment is the most common complication of stroke; it was measured by FMA quantitatively. The scale is divided into 5 domains; sensory & motor function, balance, joint range of motion and joint pain. Each domain has a scale of 0 to 2 score while the total scoring of the scale is 226 score.

CONTACTS AND LOCATIONS:
Overall Officials: IMRAN AMJAD, PhD, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Baqir, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No